CLINICAL TRIAL: NCT00257972
Title: Efficacy of Aripiprazole in Combination With Valproate or Lithium in the Treatment of Mania in Patients With Bipolar I Disorder Partially Nonresponsive to Valproate or Lithium Monotherapy
Brief Title: Study of Aripiprazole in Patients With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-134
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2008-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Mania
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The purpose of this research study is to compare the efficacy of aripiprazole with placebo in combination with lithium or valproate monotherapy, in the treatment of bipolar I patients with manic or mixed episodes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bipolar I disorder, manic or mixed episode

Exclusion Criteria:

* First manic or mixed episode
* Allergic, intolerant, or unresponsive to lithium and valproate or to aripiprazole
* Participation in a previous clinical trial within the past month or ever participated in a trial with aripiprazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in a mania rating scale

SECONDARY OUTCOMES:
Response rate and Clinical Global Impression Scale at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (90):
- United States (20):
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Riverside, California
  - Local Institution, Deerfield Beach, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, Maitland, Florida
  - Local Institution, Hoffman Estates, Illinois
  - Local Institution, Oak Brook, Illinois
  - Local Institution, Newton, Kansas
  - Local Institution, Newton, Massachusetts
  - Local Institution, New York, New York
  - Local Institution, Staten Island, New York
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Dayton, Ohio
  - Local Institution, Media, Pennsylvania
  - Local Institution, Norristown, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, Memphis, Tennessee
  - Local Institution, Austin, Texas
  - Local Institution, Bellevue, Washington
- Local Institution, Epping, Victoria, Australia
- Bulgaria (3):
  - Local Institution, Rousse
  - Local Institution, Sofia
  - Local Institution, Varna
- Czechia (4):
  - Local Institution, Brno-Bohunice
  - Local Institution, Hradec Králové
  - Local Institution, Opava
  - Local Institution, Prague
- Estonia (5):
  - Local Institution, Pärnu
  - Local Institution, Tallinn
  - Local Institution, Tartu
  - Local Institution, Viljandi Maakond
  - Local Institution, Voru Maakond
- France (10):
  - Local Institution, Bordeaux
  - Local Institution, Dole
  - Local Institution, Grenoble
  - Local Institution, Jonzac
  - Local Institution, La Rochelle
  - Local Institution, Limoges
  - Local Institution, Marseille
  - Local Institution, Nîmes
  - Local Institution, Pessac
  - Local Institution, Rennes
- Germany (5):
  - Local Institution, Berlin
  - Local Institution, Jena
  - Local Institution, Magdeburg
  - Local Institution, Meunchen
  - Local Institution, Westersted
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Gyula
  - Local Institution, Kecskemét
  - Local Institution, Nagykálló
- Italy (8):
  - Local Institution, Bassano del Grappa
  - Local Institution, Cagliari
  - Local Institution, Florence
  - Local Institution, Pisa
  - Local Institution, Roma
  - Local Institution, Sassari
  - Local Institution, Trieste
  - Local Institution, Voghera -Pavia
- Netherlands (2):
  - Local Institution, Retranchement
  - Local Institution, Zaandam
- Poland (6):
  - Local Institution, Choroszcz
  - Local Institution, Kościan
  - Local Institution, Krakow
  - Local Institution, Poznan
  - Local Institution, Torun
  - Local Institution, Tuszyn
- Local Institution, Lisbon, Portugal
- Russia (4):
  - Local Institution, Leningrad Region
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Smolensk
- South Africa (7):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Westdene, Free State
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Vereeniging, Gauteng
  - Local Institution, Welkom, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Observatory, Western Cape
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Valencia
  - Local Institution, Vitoria-Gasteiz
- Local Institution, Herisau, Switzerland
- United Kingdom (5):
  - Local Institution, Glasgow, Dumbartonshire
  - Local Institution, London, Greater London
  - Local Institution, Burnley, Lancashire
  - Local Institution, South Wales, Mid Glamorgan
  - Local Institution, Surbiton, Middlesex

REFERENCES:
- [Background] Vieta E, T'joen C, McQuade RD, Carson WH Jr, Marcus RN, Sanchez R, Owen R, Nameche L. Efficacy of adjunctive aripiprazole to either valproate or lithium in bipolar mania patients partially nonresponsive to valproate/lithium monotherapy: a placebo-controlled study. Am J Psychiatry. 2008 Oct;165(10):1316-25. doi: 10.1176/appi.ajp.2008.07101560. Epub 2008 Apr 1. PMID 18381903
- [Derived] Vieta E, Owen R, Baudelet C, McQuade RD, Sanchez R, Marcus RN. Assessment of safety, tolerability and effectiveness of adjunctive aripiprazole to lithium/valproate in bipolar mania: a 46-week, open-label extension following a 6-week double-blind study. Curr Med Res Opin. 2010 Jun;26(6):1485-96. doi: 10.1185/03007991003779380. PMID 20429835